CLINICAL TRIAL: NCT05841264
Title: Comparison Between Children Growth Chart Parameters and Their Abnormality Associated Risk Factors in Assiut Governorate
Brief Title: Growth Chart Parameters, Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariana Noss Abdo Abdelmalak, Principal Investigator, Assiut University
Other Study IDs: Growth chart, Risk factors
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Growth Disorders
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- children's in urban area: children's in this have good socioeconomic state, small family number, good hygiene
  Interventions: Behavioral: good feeding, cleaning
- children in rural area: children's in this have bad socioeconomic state, large family number, bad hygiene
  Interventions: Behavioral: good feeding, cleaning
- children in semi urban area: children's in this have bad socioeconomic state, small family number, bad hygiene
  Interventions: Behavioral: good feeding, cleaning

INTERVENTIONS:
Behavioral: good feeding, cleaning — taking healthy food which contain minerals, vitamins essential for normal growth

SUMMARY:
comparison between growth chart parameters and different risk factors which can cause abnormal growth chart parameter

DETAILED DESCRIPTION:
Infant growth is defined as a positive change in body size over a period of time, and it is a sensitive predictor of an individuals' health. An inappropriate growth pattern indicates nutritional disorders, chronic and infectious diseases in infants. Early growth rate is related to adulthood health, such that it is important to develop the concept of appropriate growth for parents, in other to detect children with abnormal growth rates, as soon as possible .Weight and height of preschool children are the most common anthropometric measurements, to investigate a child's growth rate. Weight is the simplest and most reliable anthropometric measurement, and may be used as an indicator of childhood infection. On the other hand, height summarizes various measures of nutritional conditions in the first two decades of a human's life. Many children younger than 5 years in developing countries are exposed to multiple risks, including poverty, malnutrition, poor health, and unstimulating home environments, which detrimentally affect their cognitive, motor, and social-emotional development.

ELIGIBILITY:
Inclusion Criteria:

* All children attending primary health care units in Assiut governorate aged from one year to five year

Exclusion Criteria:

* 1. congenital anomalies 2. chronic diseases (D.M , thyroid dysfunction)

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children living in different areas have low incomes, high fertility, and provide poor care form their parents different socioeconomic state, different type of food
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
comparison of growth and development of children in different areas in Assiut governorate | through study completion, an average of 1 year
  by using WHO growth chart for weight and height parameter, if child weight and height in normal average or not

SECONDARY OUTCOMES:
factors affecting growth and development of children in different areas in Assiut governorate | through study completion, an average of 1 year
  questionnaire about different factors that can affect child growth

IPD SHARING:
Plan to Share IPD: Undecided